CLINICAL TRIAL: NCT00390351
Title: Diagnosis of Non-Melanoma Skin Cancer With Optical Coherence Tomography
Brief Title: Investigate the Diagnostic Value and Possibilities of OCT in Non-Melanoma Skin Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Other Study IDs: oct-MM-2005; Grant # BIOPHOT 26-02-0020
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2006-10-19 (Estimated); Status verified 2006-10

CONDITIONS: Skin Neoplasms
Keywords: Optical coherence tomography
MeSH Terms: conditions — Skin Neoplasms | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Device: optical coherence tomography

SUMMARY:
We will do systematic and functional assessment of non-melanoma skin cancer including precancerous lesions by OCT imaging and other diagnostic methods. The systematic assessment will be comparison of clinical diagnosis, histopathology, OCT images, spectrophotometry and high frequency ultrasound of non-melanoma skin cancer Functional exploration of non-melanoma skin cancer is done with Doppler-OCT and polarization-sensitive-OCT.

DETAILED DESCRIPTION:
Optimal management of skin malignancies relies on early and accurate diagnosis. The reference standard in skin cancer is biopsy and histopathological assessment from a clinical suspicious skin lesion. The clinical diagnosis of skin cancer has sensitivity ranging from 50% to 90 % and specificity around 70% to 80% depending on the population studied and the experience of the clinician.

A rapid, non-invasive technique that could be used for characterization of skin lesions prior to biopsy would be valuable. In some patients with multiple, recurrent skin tumours the need for numerous biopsies in the same area is problematic, both cosmetically and diagnostically, as the cancer can be hidden under scar tissue.

The biopsy has several weaknesses: The biopsy must be done exactly in the tumour, and it does not delineate the tumour borders. Biopsy from skin is in general easy, but there are problematic places such as the T-zone in the face, the eyelids and the ears. Notably these places are areas where most types of skin cancer exhibit aggressive, invasive growth and have a high recurrence rate.

OCT is a novel, non-invasive optical imaging technology. It can provide cross-sectional tomographic images of tissue pathology in situ and in real time, without the need for excision and processing of specimens, as in conventional histopathology. OCT uses harmless, infrared light to create high-resolution images of tissue. OCT provides cross-sectional images of structures below the tissue surface in analogy to histopathology. Hence OCT can function as an "optical biopsy" providing images of tissue structure on the micron scale. For example, OCT could be used where standard excisional biopsy is hazardous or impossible, and OCT could reduce sampling errors associated with excisional biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 years with primary non-melanoma skin cancer NMSC or precancerous lesions from the Dermatology Department, and the Plastic Surgery Department at Roskilde Hospital, and from office based dermatologist in Roskilde County. Patients will only be recruited after informed consent.

Exclusion Criteria:

* Pregnancy.
* To avoid the potential bias of scar tissue in the OCT images we will not include OCT images from recurrent NMSC in this study.
* Patients will be excluded from the study if they are not able to give an informed consent. Staff from the Dermatology, Internal Medicine and Plastic Surgery Departments at RAS cannot be included in the phase I/phase 2 study.
* Gender: both
* Age limits: 18- no max

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-02; Study Completion 2008-07

CONTACTS AND LOCATIONS:
Overall Officials: Mette Mogensen, MD, Principal Investigator — Dept. of Dermatology, Roskilde Hospital; Gregor BE Jemec, MD, DMSc, Study Director — Dept. of Dermatology, Roskilde Hospital
Locations (2):
- Denmark (2):
  - Roskilde Hospital, Roskilde, Roskilde
  - Dept. of Dermatology, Copenhagen University, Dk-4000 Roskilde